CLINICAL TRIAL: NCT04410263
Title: Microbiota in COVID-19 Patients for Future Therapeutic and Preventive Approaches
Acronym: MICRO-COV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00646
Record Dates: First submitted 2020-05-18; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Corona Virus Infection; ARDS; Coinfection
Keywords: COVID 19; SARS Cov2; Coinfection
MeSH Terms: conditions — Coronavirus Infections; Coinfection; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-positive ICU patients: The collective of COVID-positive patients on the ICU
  Interventions: Diagnostic Test: Sampling (EDTA blood, pharyngeal and nose swabs, bronchoalveolar lavage ,urine)

INTERVENTIONS:
Diagnostic Test: Sampling (EDTA blood, pharyngeal and nose swabs, bronchoalveolar lavage ,urine) — Most data and part of the biological material required for addressing the research questions in this project are generated in the treatment of the patients. The following data and samples are collected specifically for this project according to the study schedule (i.e. extra sampling or additional questioning):
  * blood samples (day 0= 40 ml EDTA, day 2= 20 ml EDTA, day 3= 30 ml EDTA, day 5=10 ml EDTA, every 5 days = 20 ml EDTA)
  * Swabs (oral +/- nasal +/- nasopharyngeal)
  * Sublingual microscopy
  Other Names: Sublingual microscopy

SUMMARY:
In light of the rapidly emerging pandemic of SARS-CoV-2 infections, the global population and health care systems are facing unprecedented challenges through the combination of transmission and the potential for severe disease. Acute respiratory distress syndrome (ARDS) has been found with unusual clinical features dominated by substantial alveolar fluid load. It is unknown whether this is primarily caused by endothelial dysfunction leading to capillary leakage or direct virus induced damage. This knowledge gap is significant because the initial balance between fluid management and circulatory support appear to be decisive. On progression of the disease, bacterial superinfection facilitated by inflammation and virus related damage, has been identified as the main factor for patient outcome, but the role of the host versus the environment microbiome remains unclear.

The overarching aim of the present research proposal is to improve therapeutic strategies in critically ill patients with ARDS due to SARS-CoV-2 infection by advancing the pathophysiological understanding of this novel disease. This research thus focuses on inflammation, microcirculatory dysfunction and superinfection, aiming to elucidate risk factors (RF) for the development of severe ARDS in SARS-CoV-2 infected patients and contribute to the rationale for therapeutic strategies. The hypotheses are that (I) the primary damage to the lung in SARS-CoV-2 ARDS is mediated through an exaggerated pro-inflammatory response causing primary endothelial dysfunction, and subsequently acting two-fold on the degradation of the lung parenchyma - through the primary cytokine response, and through recruitment of the inflammatory-monocyte-lymphocyte-neutrophil axis. The pronounced inflammation and primary damage to the lung disrupts the pulmonary microbiome, leading secondarily to pulmonary superinfections. (II) Pulmonary bacterial superinfections are a significant cause of morbidity and mortality in COVID-19 patients. Pathogen colonization main Risk Factor for lower respiratory tract infections. To establish colonization, pathogens have to interact with the local microbiota (a.k.a. microbiome) and certain microbiome profiles will be more resistant to pathogen invasion. Finally, (III) Handheld devices used in clinical routine are a potential reservoir and carrier of both, SARS-CoV-2, as well as bacteria causing nosocomial pneumonia.

DETAILED DESCRIPTION:
In December 2019, severe pneumonia cases were reported in relation to the Huanan Seafood Wholesale Market in Wuhan, China. Four months and more than thousand deaths later, the responsible pathogen of the largest and most critical global health emergency in the last 100 years is known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The Coronavirus Disease 2019 (COVID-19) is characterized as a transmittable disease with a long incubation period of between 7 and 14 days. In around 10% of cases a severe disease course is observed. While predisposing factors such as older age, chronic arterial hypertension, diabetes, as well as other comorbidities have been described, little is known about the pathophysiological mechanism, which induce acute lung failure, coupled to the often-appearing heart, kidney and vascular injury pathognomonic for the deadly course of this disease.

The alveolar exudative and interstitial inflammation impairing alveolo-capillary gas exchange described in relation to SARS-CoV-2 complies with the definition of acute respiratory distress syndrome (ARDS). The pathophysiological mechanics behind this injury to the lung have been best described in bacterial sepsis induced ARDS, and are mainly induced by the extravasation of neutrophil granulocytes from the capillary vasculature into the lung. One of the main mediators of neutrophil extravasation is the degeneration of the endothelial surface layer, namely the glycocalyx, induced by endotoxin-activated heparan sulfate. The thinning and destructuration of the glycocalyx reveal hidden endothelial surface adhesion molecules like VCAM-1 and ICAM-1. The thereby increased adhesion of Neutrophils coupled to the inflammatory cytokine mediated dis-placement of VE-cadherin to the insides of the endothelial cells, loosening the endothelial tight junctions, allows for an increased extravasation of neutrophils and diffusion of protein-rich fluid into the interstitium. The thereby created milieu induces neutrophil granulocytes activation and degranulation, and provokes the release of toxic mediators that destroy the alveolar epithelium and produce further immunocytokines, induce a cytokine storm and augment neutrophil recruitment. Finally the aggregation of the inactivated pulmonary surfactant by the protein rich edema con-joined with the degenerated type 1 alveolar epithelial cells and the hyaline membrane covered, de-nuded alveolar basement membrane disrupt the gas exchange capacity of the alveolo-capilar membrane, impairing blood oxygenation and decarboxylation.

In contrast to bacterial-induced ARDS, viral agents causing ARDS mainly reach the alveolar epithelium through viral transport from the nasopharynx, from the upper to the lower respiratory tract. In viral infections, the damage to the lung is primarily caused by a direct viral invasion of type 1 and 2 pneumocytes. This causes the accumulation of protein-rich edema in a two-fold fashion by disabling the ENaC channels, mainly responsible for the decongestion of the alveolar room through osmotic gradient creation, and by breaching the physio-chemical barrier established by the pneumocytes. Albeit the effect of alveolar barrier disruption by means of vascular endothelial dysfunction being reduced in contrast to bacterial sepsis, with the ARDS advancing, both the endothelium and epithelium secrete chemotactors to attract macrophages and neutrophils to the inflamed lung, which in analogy to bacterial ARDS induce a secondary damage to the lung as already described. However point to an exaggerated initial capillary leak as compared to other forms of ARDS, which strongly suggests endothelial dysfunction as a primary mechanism.

Endothelial cell damage may be assessed using both glycocalyx degradation products such as syndecan-1, heparan sulfate, and VE-cadherins and direct visualization of red blood cell flow properties within the capillaries via handheld vital microscopy (HVM) employing the dark field microscopy technique. Recent advances in the investiagtors group have enabled the accurate differentiation of modes of microcirculatory failure by quantification of the microcirculatory diffusion and convection capacity. From a global perspective, the alveolar leakage has previously been quantified using transpulmonary thermodilution. These tools provide the optimal prerequisites to specifically detect (glycocalyx degradation products in the alveolar lavage fluid) and quantify (transpulmonary thermodilution) endothelial cell damage in the lung during ARDS caused by SARS-CoV-2 infection. Further, approximately 20% of critically ill patients suffering from ARDS due to SARS-CoV-2 infection have been described in preliminary reports to develop severe systemic inflammatory response and circulatory shock. In these patients, the relation between alveolar endothelial cell damage and systemic endothelial cell damage is of central interest and may be assessed by concomitant sublingual HVM measurement.

Following the viral and inflammatory mediated lung damage as the initial trigger for ARDS, the further deterioration of the lung function may mainly depend upon superinfection. Bacterial and fungal superinfection has been described as mainly responsible for morbidity and mortality in mid- to late-phase viral ARDS during similar pandemics, such as the Spanish Flu in 1918. In the current outbreak in China, presence of bacterial and fungal superinfections was found in 10 to 30%. Superinfection seemed to represent a major risk factor for mortality in the COVID-19 patients. Albeit being unclear if detection of bacterial and fungal superinfection has a clinical and therapeutic relevance, several authors advocate empirical antibiotic treatment targeting mainly S. aureus and S. pneumonia.

Not only is the stratification of risk associated with bacterial and fungal superinfections relevant to the assessment of severity of disease progression, but the question remains to be assessed to which degree the presence of nosocomial pathogen transmission during pandemics exists and is responsible for morbidity and mortality in hospitalized patients. Infection prevention measures, such as standard and isolation precautions, are intended to prevent the nosocomial transmission of pathogens in healthcare settings. These measures include hand hygiene, the use of personal protective equipment (PPE) (e.g. isolation gowns, gloves, masks, respirators, eye protection), and environmental measures - such as the cleaning and disinfecting of surfaces and medical equipment and instruments. Yet, mobile devices, such as private and professional mo-bile phones, have largely been unaddressed by such guidelines. These devices may play an important role in indirect contact transmission. That is, when a contaminated intermediate object is involved in the transfer of an infectious pathogen between two individuals.

Current evidence, although limited, has shown an increased viability of SARS-CoV-2 on plastic and stainless steel, materials frequently employed on mobile devices and protective covers, of up to 72 hours. Albeit incorrect hand hygiene, lack of personal protective equipment and other hygienic routine mistakes are the most obvious vectors of nosocomial pathogens, mobile phones and other handheld devices have been found to be insufficiently disinfected, allowing pathogen colonization, of which S. aureus is the most frequent. This is aggravated by the fact that healthcare providers touched mobile objects, including mobile phones, on average once every 6.9 seconds and touched their own body or face every 40 seconds. This was accompanied by an extremely low adherence to hand hygiene protocols prior to colonization and infection events. These findings underline the potential of mobile devices, to act as vectors of transmission of pathogens to both patients and healthcare providers.

In combating viral infections, the innate immune defense recognizes viral infection mainly through binding of pathogen associated molecular patterns (PAMPs) to pathogen-recognition receptors (PRRs). The expression cascade induced by these receptor bindings stimulates the Interferon (IFN) Type I and III pathway. The recruitment of the inflammatory monocyte-macrophage-neutrophil axis by the IFN I pathway is essential in the fight against most viral infections. Neverthe-less, viruses such as the Influenza A virus are capable of evading the IFN type I and III inception, by moving their replication machinery into the cell nucleus thus evading the cytoplasmically located PRRs or inactivating interferon mRNAs through proteins. The IFN I pathway can act two-fold in these viruses; on one side it may mediate initial action against the virus reducing maximal reached titers, on the other hand, under certain circumstances it can nevertheless pathologically overex-press inducing a cytokine storm and increasing damage to the lung parenchyma.

SARS-CoV and SARS-CoV-2 are positive-strand RNA viruses, which penetrate the cellular wall of the infected cells by ACE-2 receptor mediated endocytosis. A onset of the IFN I pathway expression may be associated with a stronger IFN II pathway activation and pro-inflammatory cytokine storm induction and consequently a more severe dysregulation of the inflammatory monocyte-macrophage system and the degree of lung immunopathological damage. The pathophysiological mechanics of this new SARS-CoV-2 induced ARDS and the systemic dysregulations it induces can only be speculated based on its predecessor SARS-CoV, and insights elucidating the unusual clinical presentation of the novel disease are desperately needed to derive an optimal treatment approach.

In summary, the mechanisms of disease severity in critically ill SARS-CoV-2 ARDS are manifold, ranging from a dysregulated inflammatory response, over the presence of bacterial and fungal superinfections to the importance of nosocomial transmission as a key targetable element in day-to-day patient care. Only a global assessment of all facets possibly responsible for the severity of dis-ease progression in COVID-19 patients, can aim to elucidate the underlying concoction.

Project Objectives The overarching aim of this research is to gain the pathophysiological understanding to improve morbidity and mortality in ARDS due to SARS-CoV-2 infection. This research thus focuses on inflammation, microcirculatory dysfunction and superinfection, aiming to elucidate risk factors for the development of severe ARDS of SARS-CoV-2 infected patients and contribute to the rationale for therapeutic strategies.

The individual working hypotheses are:

1. The primary damage to the lung in SARS-CoV-2 ARDS is thought to be mediated by an exaggerated pro-inflammatory response causing primary endothelial dysfunction, and subsequently acting two-fold on the degradation of the lung parenchyma, through the primary cytokine response, and through recruitment of the inflammatory-monocyte-lymphocyte-neutrophil axis. The pronounced inflammation and primary damage to the lung disrupt the pulmonary microbiome, leading secondarily to pulmonary superinfections.
2. Pulmonary bacterial superinfections (i.e., S. pneumoniae, S. aureus, P. aeruginosa and others) are a significant cause of morbidity and mortality in COVID-19 patients. Pathogen colonization in the upper airways is a prerequisite and the main risk factor for lower respiratory tract infections. To establish colonization, pathogens have to interact with the local microbiota (a.k.a. microbiome) and certain microbiome profiles will be more resistant to pathogen invasion.
3. Handheld devices used in clinical routine are a carrier of both, SARS-CoV-2, as well as bacteria causing nosocomial pneumonia, making them a potential reservoir for indirect contact transmission. A targeted infection prevention intervention can reduce this contamination and thereby reduce the risk of nosocomial transmission.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years on day of inclusion
* SARS-CoV-2 infection confirmed according to WHO guidelines
* Hospitalization in intensive care unit for severe ARDS
* Confirmation of an independent doctor to safeguard the interests of the patient

Exclusion Criteria:

• Visible opposition to participate in the research project, expressed either verbally or through behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID 19 patients admitted to the intensive care unit of the University Hospital Zurich
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of pro-inflammatory response over the ICU stay as a causative for primary endothelial dysfunction | Admission, on day 0, day 1, day 2 , day 3, day 5, every 5 days up to 1 year
  Daily recorded Vitals and Inflammatory Response will be analyzed by means of multivariable mixed effect models analysis and generalized linear models, with corrections for time and randomness. To account for the different units of measure we will standardize all values to an absolute measure by means of the z-score.
  The following variables will be considered:
  Respiratory values, Vital signs, Haemodynamic monitoring, Microcirculation, Inflammatory values, Hematology: T-cells CD3, 4 and 6 Chemistry: Inflammatory Cytokines and Biomarkers:CRP, PCT, MR-ProADM, IFN-1, IFN-γ, TNF-α/β, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, MIG, RANTES, MCP-1, IP-10, PD1, PD-L1 Lipid-pannel3: LDL, HDL, Cholesterol, Triglyceride Other: HLA DR/DQ TBS, Swabs, sublingual nonnvasive microscopy
Time-to-event "pulmonary bacterial superinfection or death" | Through study completion, an average of 30 days
  COX proportional hazards model and generalized mixed effect models assessing the effect of positive bacterial infection on mortality. Correction for time and randomness (multiple sampling).
  Super infection will be defined as a positive bacterial/ fungal sample (Bood cultures, BAL, TBS, Swabs, Urine)
Positive bacteria and/ or SARS-CoV-2 cultures on handheld devices used in clinical routine and correlation to the adherence to disinfection protocols | Through study completion, an average of 30 days
  Mobile devices will be swabed for bacterial and viral contamination, simultaneously adherence of the user to disinfection protocols will be assessed.

SECONDARY OUTCOMES:
Life Quality after COVID-19 Infection | follow up 30 + 90 days and 1 year after discharge
  SF 36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Brugger, SB, Principal Investigator — USZ; Philipp K Buehler, PB, Study Chair — USZ
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strickler NS, Hofmaenner DA, Schuepbach RA, Scheier TC, Buehler PK, Takala J, Brugger SD, Frey PM. Use of carbon dioxide production to detect bacterial superinfections in mechanically ventilated patients with acute respiratory distress syndrome: an exploratory prospective cohort study. BMJ Open Respir Res. 2025 Aug 28;12(1):e002760. doi: 10.1136/bmjresp-2024-002760. PMID 40876958
- [Derived] Busnadiego I, Abela IA, Frey PM, Hofmaenner DA, Scheier TC, Schuepbach RA, Buehler PK, Brugger SD, Hale BG. Critically ill COVID-19 patients with neutralizing autoantibodies against type I interferons have increased risk of herpesvirus disease. PLoS Biol. 2022 Jul 5;20(7):e3001709. doi: 10.1371/journal.pbio.3001709. eCollection 2022 Jul. PMID 35788562